CLINICAL TRIAL: NCT06549049
Title: A Randomized, Controlled Trial of a Modified Sleep and Circadian Intervention for Veterans With PTSD: Advancing Psychosocial Rehabilitation Through Sleep Health
Brief Title: A Transdiagnostic Sleep Health Intervention for Veterans With PTSD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D4796-R
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Stress Disorders, Post-Traumatic; Sleep Initiation and Maintenance Disorders
Keywords: Insomnia; Posttraumatic stress disorder; Veterans; Nightmares; Psychotherapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: The study involves a randomized, controlled, single-blind trial to evaluate the effectiveness of TranS-C modified for Veterans with PTSD (TSC-PTSD) in male and female Veterans who are enrolled in primary and/or mental health care in the VA system. Study treatment will be implemented remotely via live video visits using a VA-approved platform. Enrolled participants will be randomly assigned to the TSC-PTSD group or to the sleep psychoeducation control (SPC) group.
Who Masked: Participant
Masking Description: This is a single-blind study. Participants will not know to which group they are assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Experimental (Experimental): Participants receiving experimental TSC-PTSD treatment.
  Interventions: Behavioral: TranS-C for PTSD
- Arm 2: Active Control (Active Comparator): Participants receiving sleep psychoeducation control.
  Interventions: Behavioral: Sleep Psychoeducation Control

INTERVENTIONS:
Behavioral: TranS-C for PTSD — The Transdiagnostic sleep and circadian intervention (TranS-C), developed by Allison Harvey, Ph.D. and Daniel Buysse, M.D., involves a patient-centered, module-based, flexibly structured approach that tackles numerous sleep disturbances using evidence-based strategies with the goal of improving sleep and related impairments in daytime functioning. It is thus well-suited for tackling sleep disturbances and the associated impairments in social, occupational and overall functioning in veterans with PTSD. The proposed study is a randomized, controlled clinical trial examining the effectiveness of a modified TranS-C intervention for veterans with PTSD. The modified approach, TranS-C for PTSD (TSC-PTSD), elevates the importance of nightmare-focused, apnea-focused, and insomnia-focused modules relative to the standard intervention, incorporates an evidence-based relaxation module, and modifies the nightmare and apnea modules based on strategies used for veterans in the VA healthcare system.
  Other Names: TSC-PTSD
  Arms: Arm 1: Experimental
Behavioral: Sleep Psychoeducation Control — Participants will receive psychoeducation about sleep.
  Other Names: SPC
  Arms: Arm 2: Active Control

SUMMARY:
Sleep disturbance is a major problem in Veterans with posttraumatic stress disorder (PTSD). This study will test a version of a sleep treatment that's been shown to be effective in the general population, with some changes to tailor it to the needs of Veterans with PTSD and sleep disturbance.

DETAILED DESCRIPTION:
Sleep disturbance in military Veterans with PTSD is a complex condition, typically characterized by insomnia and nightmares, and frequently accompanied by comorbid obstructive sleep apnea. Each of these problems are shown to influence the others, contributing to a complex sleep disturbance with profound impacts on daytime functioning and quality of life. A vicious cycle in which nighttime disturbances impact daytime functioning, and vice versa, often ensues. Addressing sleep disturbance in Veterans with PTSD therefore requires a multipronged approach that is tailored to each Veterans' constellation of symptoms and each Veterans' goals for sleep health. The Transdiagnostic sleep and circadian intervention (TranS-C), developed by sleep researchers Allison Harvey, Ph.D. and Daniel Buysse, M.D., involves a patient-centered, module-based, flexibly structured approach that tackles numerous sleep disturbances using evidence-based strategies with the overall goal of improving sleep and improving sleep-related impairments in daytime functioning. It is thus well-suited for tackling sleep disturbances and the associated impairments in social, occupational and overall functioning in Veterans with PTSD. The proposed study is a randomized, controlled clinical trial examining the effectiveness of a modified TranS-C intervention for Veterans with PTSD. The modified approach, referred to as TranS-C for PTSD (TSC-PTSD) elevates the importance of nightmare-focused, apnea-focused, and insomnia-focused modules relative to the standard intervention, incorporates an evidence-based relaxation module, and modifies the nightmare and apnea modules based on strategies used for Veterans in the VA healthcare system. The study will administer TSC-PTSD remotely to Veterans in their homes using a VA-approved video-conferencing platform. The study will recruit male and female U.S. military Veterans aged 18 and above throughout California and compare change in a comprehensive measure of daytime functioning and change in insomnia, nightmare and overall PTSD symptoms in participants randomized to the active intervention TSC-PTSD vs. participants randomized to a sleep psychoeducation control (SPC) intervention. The widely used and validated World Health Organization Disability Assessment Schedule (WHODAS) will serve as the primary outcome measure. The Insomnia Severity Index (ISI) and the Clinician-Administered PTSD Scale (CAPS) will be used to measure secondary outcomes. Eligible participants will have an insomnia diagnosis, a PTSD diagnosis (or moderate symptoms of PTSD in the absence of a full diagnosis), and clinically significant nightmares based on gold-standard clinician-administered interviews. All participants will complete baseline surveys related to daytime functioning and sleep-related symptoms prior to treatment initiation, and will complete these surveys again in week 5, and at the end of treatment. For additional high-resolution data on sleep patterns, all participants will record sleep-related information, including nightmare occurrence and severity, in the morning and at bedtime using a Veteran-tested and user-friendly sleep diary mobile app. Participants will also complete the clinical interview and self-report surveys at 3-month and 6-month follow-up, to assess the durability of treatment effects. The duration of TSC-PTSD may vary between a minimum of 8 and a maximum of 12 sessions and the psychoeducation control protocol will involve 10 sessions. The hypotheses are: 1) subjects randomized to TSC-PTSD will demonstrate greater improvement in WHODAS score relative to SPC from baseline to post-treatment; 2) subjects randomized to TSC-PTSD will demonstrate greater improvements in insomnia, nightmares and PTSD symptoms as demonstrated by improvements in the ISI, CAPS distressing dreams score, and CAPS total score relative to SPC from baseline to post-treatment; and 3) subjects randomized to TSC-PTSD will demonstrate greater sustained improvement in functional and clinical outcomes at 3-month and 6-month follow-up relative to SPC, and improvements in WHODAS score will be mediated by improvements in ISI, nightmares and TranS-C indicators of sleep health in both study groups. Findings in support of the investigators' hypotheses will provide a vital new tool for advancing rehabilitation in U.S. military Veterans with PTSD.

ELIGIBILITY:
Inclusion Criteria:

* U.S. Military Veteran aged 18 and above engaged in VA primary and/or mental health care
* CAPS 5 PTSD diagnosis; or CAPS 5 score >=25 in the absence of full criteria
* SCID Insomnia Disorder diagnosis, supported by ISI score >=10
* CAPS-IV nightmare score >=4
* Sleep-related functional impairment based on a WHODAS score >=32
* Willingness to engage in 8-12 sessions of treatment to address their sleep disturbance

Exclusion Criteria:

* Current cognitive problems, active psychosis or mania, or other mental/cognitive conditions such as moderate to severe neurodegenerative disease that would render the participant unable to connect to videoconferencing platform, engage in remote psychotherapy, or communicate using the required VA secure email platform
* No access to reliable internet service connected to a computer, iPad or similar device (telephone not adequate)
* Inability or unwillingness to use a VA-approved videoconferencing platform and VA secure email;
* Current engagement in a sleep-focused psychotherapy, or plan to start a sleep-focused psychotherapy in the next 3 months. Sleep-focused psychotherapies include, but are not limited to, CBT-I, BBT-I, and IRT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
World Health Organization Disability Assessment Schedule (WHODAS) | Week 0, Week 5, Post-Treatment, 3-Month Follow-Up, 6-Month Follow-Up
  The WHODAS is a validated, comprehensive measure of health-related disability.

SECONDARY OUTCOMES:
Insomnia Severity Index (ISI) | Week 0, Week 5, Post-Treatment, 3-Month Follow-Up, 6-Month Follow-Up
  The ISI will be used to measure change in severity of insomnia symptoms.
Clinician-Administered PTSD Scale for DSM-4 Distressing Dream Score (CAPS-4 Nightmare Item) | Week 0, Week 5, Post-Treatment, 3-Month Follow-Up, 6-Month Follow-Up
  The CAPS-IV Nightmare Item will be used to measure change in nightmare symptoms.
Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) | Week 0, Post-Treatment, 3-Month Follow-Up, 6-Month Follow-Up
  The CAPS-5 will be used to measure change in overall PTSD symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Richards, MD MPH, Principal Investigator — San Francisco VA Medical Center, San Francisco, CA
Locations (1):
- San Francisco VA Medical Center, San Francisco, CA, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Richards Lab website — https://richardslab.ucsf.edu/